CLINICAL TRIAL: NCT02458495
Title: Leveraging Patient Portals to Improve Medication Adherence in Type 2 Diabetes
Brief Title: The Diabetes Medication Adherence Promotion Intervention Trial
Acronym: Diabetes MAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Chandra Osborn, Assistant Professor of Medicine & Biomedical Informatics, Co-Director for CHBHE, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: K01DK087894 (NIH); K01DK087894 (NIH)
Record Dates: First submitted 2015-05-26; First posted 2015-06-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Internet; Mobile Health; Hemoglobin A, Glycosylated; Medication Adherence; Psychological Theory
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care Control Group (No Intervention): Participants will be granted access to a generic Diabetes website. Participants will complete the same eligibility and baseline self-report as the intervention group. The 1 month and 3 month self-report survey will omit mention of the Diabetes MAP website and will reference the generic diabetes website.
  Participants will be provided with access to a generic Diabetes website. Participants will complete the same eligibility, baseline and self-report surveys as the intervention group.
- Diabetes MAP Intervention Group (Experimental): Participants will be granted access to the Diabetes MAP website. Participants will complete the same eligibility and baseline self-report as the control group. The 1 month and 3 month self-report will refer to the Diabetes MAP website specifically.
  Interventions: Behavioral: Diabetes MAP Intervention

INTERVENTIONS:
Behavioral: Diabetes MAP Intervention
  Arms: Diabetes MAP Intervention Group

SUMMARY:
A significant percentage of persons with diabetes fail to properly take their prescribed oral hypoglycemic agents (OHA) and insulin. Non-adherence to medications among diabetes patients is associated with poor health outcomes including suboptimal glycemic control, diabetes-related complications, elevated health costs and increased risk of hospitalization and mortality. Given the substantial impact of non-compliance on the health of patients, prior studies have sought to draw links between medication adherence and patient factors.

Research shows that web-based interventions that support patients' medication-related knowledge, motivation and skills effectively improve compliance.

The purpose of this study is to evaluate the impact of a patient web portal (PWP)-delivered medication adherence promotion intervention on medication adherence and glycemic control among patients with type 2 diabetes (T2DM). The intervention aims to (1) increase self-reported adherence to glucose lowering agents (GLAs) and (2) improve diabetes health outcomes (decreased HbA1c) by increasing patients' medication adherence-related knowledge, motivation and skills.

This research will greatly enhance the investigators' understanding of medicine compliance and the factors that effectively improve adherence among high-risk patients with diabetes. Knowledge gained from this work may inform future internet-based patient portals that support disease management and medication adherence more broadly.

DETAILED DESCRIPTION:
[Background]

Medication non-adherence is a major public health issue for patients with diabetes. Approximately one third of patients with T2DM are non-compliant with their diabetes medication. This is problematic since suboptimal medication adherence has been shown to contribute to inferior glycemic control, increased healthcare costs, hospitalization and premature death. The aforementioned ramifications of nonadherence to chronic medication are a product of barriers to diabetes self-care behavior including patient-related factors associated with glycemic control. Dr. Chandra Osborn and colleagues have identified targetable patient factors related to patients' medication-adherence related knowledge (e.g., information about medication purpose and dosage), motivation (e.g., awareness of medication benefits, social support for adherence) and self-efficacy or skills (e.g., ability to remember dosages and obtain refills). Said factors map onto the Information-Motivation-Behavioral skills (IMB) model, which has informed effective adherence promotion interventions among individuals with other chronic illnesses and may have utility in promoting medication adherence among patients with T2DM.

Intervention content will be informed by a validated theory of medication adherence. Interventions are seldom informed by empirically established theories. This is problematic since theory-based interventions (i.e., interventions that draw upon theories that are relevant to the target population) have proven to be more effective than atheoretical interventions. Few published intervention studies specifically address medication adherence among adults with T2DM and of these limited studies, only one is grounded in theory. The study's web-based intervention is driven from the aforementioned IMB model of adherence. This model incorporates central components of other theoretical models and has been validated in cross-sectional and intervention research among patients with acquired illnesses. Furthermore, recent empirical findings indicate the IMB model's success in predicting outcomes in our target T2DM population. Thus, it is reasonable to believe an intervention (i.e., Diabetes MAP) that delivers IMB model-based content to a T2DM population may successfully improve medication compliance.

Patient web portal (PWP)-delivered medication adherence promotion interventions are a practical tool for relaying health-related information and resources. The magnitude of the consequences associated with nonadherence to chronic medications makes web-based interventions imperative as they aim to reduce the impact of barriers to medication-taking practices. While there are few medication adherence promotion interventions specifically designed for patients with T2DM, the literature suggests barriers to medication adherence practices may be reduced with the use of interactive behavior change technologies (IBCT) that provide patients with access to resources, web tools and health knowledge. While there can be limitations to patient websites (e.g., poor design), the usability of the web-based health intervention Diabetes MAP has been previously evaluated in relation to ease of interaction and accessibility to individually-tailored components aimed at increasing diabetes-related knowledge, motivations and skills. This study aims to leverage the use of Diabetes MAP to help T2DM patients overcome barriers to self-care and promote medication adherence behavior and improve diabetes outcomes.

Personality measures may moderate adherence and effectiveness of a PWP-delivered intervention. In an attempt to broaden our understanding of self-care behavior, the study implements an additional instrument, the Mindful Attention Awareness Scale (MAAS), to obtain a personality measure of mindfulness. Mindfulness is a psychological construct of Buddhist origin that draws together deliberate attention to moment-to-moment occurrences and the cultivation of knowledge, positive emotions and ethical behavior. The MAAS is a validated 15-item scale designed to measure an individual's awareness and ability to attend to what is occurring in the present moment. Studies indicate that the quality of mindfulness targeted by the MAAS is related to, and predictive of, certain self-regulation and well-being constructs. More specifically, mindfulness has been linked to increased subjective well-being, reduced psychological symptoms and reactivity, and improved behavioral regulation, all of which may be correlated with self-care behavior and better decision making regarding health (i.e., diet, exercise). Therefore, study participants with high baseline levels of self-awareness may draw even greater benefits from use of the Diabetes MAP website and therefore display greater medication adherence and lower A1c levels than those scoring lower on the MAAS.

[Study Objective/Aim]

The goal of this research is to evaluate a web-based medication adherence promotion intervention that uses patient-specific information (e.g., diabetes medication, survey responses) to deliver tailored content via the Diabetes MAP website to adults with T2DM.

The specific aim is to evaluate the ability of an existing PWP-delivered medication adherence promotion intervention (Diabetes MAP) to improve medication adherence and glycemic control among patient participants with T2DM. Investigators will randomly allocate patients to a treatment (website intervention or no intervention) and subsequently test the website's ability to increase self-reported adherence to glucose lowering agents (GLAs) and improve diabetes health outcomes as demonstrated by lowered HbA1c levels.

[Significance]

This project evaluates the effect of the PWP-delivered medication adherence promotion intervention, Diabetes MAP, on patient adherence to glucose lowering agents (GLAs) and patient HbA1c. The study serves to fill the gap in the current literature by focusing on the power of interactive and individually-tailored technology to support medication adherence and the subsequent health benefits that arise when T2DM patients properly adhere to their prescribed medical regimen. In addition to reducing personal costs (e.g., hospitalization, mortality, healthcare fees), improving medication adherence among T2DM patients may benefit society by reducing the burden said individuals' health status places on the broader population. Ultimately, the tools and techniques utilized and the data collected from this study will provide insight for future studies that may seek to utilize web-based interventions to reach and impact medically afflicted individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older (to be confirmed by electronic health record)
* Individuals who have received a diagnosis for type 2 diabetes mellitus (T2DM)
* Enrolled as a patient in the Vanderbilt APPC or the Eskind Diabetes Clinic
* Registered My Health at Vanderbilt user
* Recent A1c of 7.0 or greater
* Individuals currently being treated with oral and/or injectable diabetes medication (to be confirmed through electronic health record)

Exclusion Criteria:

* Non-English speakers (determined by a trained research assistant)
* Individuals with a severe hearing or visual impairment (determined subjectively by a trained research assistant)
* Individuals with delirium or a severe cognitive impairment (determined by a lack of orientation to person, place, and time)
* Individuals who report a caregiver administers their diabetes medications
* Individuals who report they do not have a mobile phone or computer with internet access
* Individuals unwilling and/or unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2015-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Glycemic control (Change in participant's HbA1c level) | Change from Baseline in HbA1c level at 3 months
  Change in participant's HbA1c level from study onset to study conslusion

SECONDARY OUTCOMES:
Number of logins, 1 month assessment | 1 month after Baseline
  Web analytics will be implored to measure participant engagement with Diabetes MAP website demonstrated by number of user logins to website between baseline and 1 month assessment
Number of logins, 3 month assessment | 3 months after Baseline
  Web analytics will be implored to measure participant engagement with Diabetes MAP website demonstrated by number of user logins to website between baseline and 3 month assessment
Time spent on website, 1 month assessment | 1 month after Baseline
  Web analytics will be implored to measure participant engagement with Diabetes MAP website demonstrated by times spent on website between baseline and 1 month assessment
Time spent on website, 3 month assessment | 3 months after Baseline
  Web analytics will be implored to measure participant engagement with Diabetes MAP website demonstrated by times spent on website between baseline and 3 month assessment

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Y Osborn, PhD, MPH, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States